CLINICAL TRIAL: NCT05037175
Title: Telehealth 2.0: Evaluating Effectiveness and Engagement Strategies for Asynchronous Texting Based Trauma Focused Therapy for PTSD
Brief Title: Telehealth 2.0: Evaluating Effectiveness and Engagement Strategies for CPT-Text for PTSD
Acronym: CPT-TEXT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); Talkspace (Industry); National Institute of Mental Health (NIMH) (NIH); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Shannon Wiltsey Stirman, PhD, Associate Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 62509; RF1MH128785 (NIH)
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Digital Mental Health; COVID-19
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CPT-Text + Incentive (Experimental): CPT-Text. CPT is a 12-session (13 text-based modules), trauma-focused, cognitive therapy that teaches clients to examine and change problematic beliefs about themselves and the world that were altered as a result of trauma. Clients can work at their own pace.
  Retention Incentive (RI). Participants will be told at baseline that they can earn discounts for other users with PTSD if they message with their therapist regularly.
  Interventions: Behavioral: CPT-Text; Behavioral: Retention Incentive
- CPT-Text + Reminder As Usual (Experimental): CPT-Text. CPT is a 12-session, trauma-focused, cognitive therapy that teaches clients to examine and change problematic beliefs about themselves and the world that were altered as a result of trauma.
  Reminder as Usual (RAU). As per Talkspace guidelines, therapists are available to client participants twice per day, five days per week. In the event a client participant has not engaged or messaged in 48 hours, therapists send a personalized message to the client participant to encourage them to re-engage.
  Interventions: Behavioral: CPT-Text; Behavioral: Reminder as Usual
- Culturally Informed Trauma Treatment (CITT) + Incentive (Active Comparator): CITT will be conducted by Talkspace therapists with a specialty in PTSD culturally informed PTSD treatment.
  Retention Incentive for other users with PTSD in subsequent months if they message with their therapist regularly.
  Interventions: Behavioral: Culturally Informed Trauma Treatment (CITT); Behavioral: Retention Incentive
- CITT+ Reminder as Usual (Active Comparator): CITT will be conducted by Talkspace therapists with a specialty in culturally informed PTSD treatment.
  Reminder as Usual (RAU). As per Talkspace guidelines, therapists are available to client participants twice per day, five days per week. In the event a client participant has not engaged or messaged in 48 hours, therapists send a personalized message to the client participant to encourage them to re-engage.
  Interventions: Behavioral: Culturally Informed Trauma Treatment (CITT); Behavioral: Reminder as Usual

INTERVENTIONS:
Behavioral: CPT-Text — CPT is a 12-session (13 modules), trauma-focused, cognitive therapy that teaches clients to examine and change problematic beliefs about themselves and the world that were altered as a result of trauma. Each session includes psychoeducation and introduction of a new skill or module, which builds on the previous information and skills. Participants will receive psychoeducation video links via Talkspace and an electronic workbook with handouts, written explanations of the concepts and activities, and CPT worksheets, which will be embedded in the platform and sent by the therapist at the appropriate point in the protocol. Therapists encourage the client to complete each module using the provided materials and assist clients in reflecting on their beliefs through Socratic questions and feedback on their worksheets. Clients work at their own pace, with therapists sending the skill or module after the client has practiced the previous one. Brief synchronous messaging sessions can be arranged
  Arms: CPT-Text + Incentive; CPT-Text + Reminder As Usual
Behavioral: Culturally Informed Trauma Treatment (CITT) — CITT will be conducted by Talkspace therapists with a specialty in PTSD treatment. Based on previous research and Talkspace's analysis of TAU and the therapists' training in culturally informed trauma treatment, it is likely CITT will include culturally informed, supportive and client-centered interventions, problem solving, and elements from EBTs such as cognitive-behavioral therapy. Brief synchronous messaging sessions can be arranged.
  Arms: CITT+ Reminder as Usual; Culturally Informed Trauma Treatment (CITT) + Incentive
Behavioral: Retention Incentive — Participants will be told at baseline that they can earn free or discounted therapy for other individuals with PTSD who are in need of financial assistance if they remain consistently engaged in treatment. If client participants do not re-engage after 24 hours from the RAU (3 days without engagement), they will receive an automated text-message reminding them to message their therapist regularly (on average, every other business day) in order to get a discount donated it to a fund that will offer free or discounted therapy to individuals with PTSD who require financial assistance. Throughout treatment, participants will be sent reminders every other week of what the incentive is and how it can be acquired, in addition to feedback about whether they are on or off track to earn the discount.
  Arms: CPT-Text + Incentive; Culturally Informed Trauma Treatment (CITT) + Incentive
Behavioral: Reminder as Usual — As per Talkspace guidelines, therapists are available to client participants twice per day, five days per week. In the event a client participant has not engaged or messaged in 48 hours, therapists send a personalized message to the client participant to encourage them to re-engage.
  Arms: CITT+ Reminder as Usual; CPT-Text + Reminder As Usual

SUMMARY:
There is a pressing need to increase capacity to treat PTSD related to or exacerbated by the COVID-19 pandemic. Texting-based therapy holds promise to increase capacity and reduce barriers to delivering evidence-based treatments (EBTs), but ongoing engagement in digital mental health interventions is low. This study will compare a texting-based EBT for PTSD to culturally-informed texting-based treatment for PTSD as usual, and it will also compare a unique incentive strategy to typical platform reminders aimed to prevent early discontinuation in therapy. This online study is open to individuals who live in 18 different states.

DETAILED DESCRIPTION:
The COVID-19 pandemic has exacerbated mental health challenges for trauma-exposed individuals due to increased isolation, insufficient capacity in the mental health workforce, and a predicted fourth wave of mental health impacts of the pandemic itself. There is a pressing need to increase treatment capacity. Digital mental health (DMH) interventions for posttraumatic stress disorder (PTSD) address well-documented barriers to traditional in-person psychotherapy or telehealth delivery of evidence-based treatments (EBTs) for PTSD, but many consumers do not remain engaged. Thus, acceptable, efficient, and engaging forms of EBTs are sorely needed, particularly for those who are less likely to access traditional psychotherapy or use online programs. Asynchronous texting therapy platforms may facilitate treatment engagement among those who seek discrete, convenient, and affordable support. In a pilot study of a texting-based format of an EBT for PTSD, Cognitive Processing Therapy (CPT-Text), CPT-Text was feasible to deliver, and clients showed substantially greater PTSD symptom improvement over a shorter time compared to text therapy as usual (TAU). A larger scale, more rigorous test is necessary. This is a randomized, Hybrid Type 1, effectiveness-implementation trial with a factorial design to compare text-based therapies for PTSD utilizing the HIPAA-compliant secure texting platform of our DMH partner, Talkspace. Participants will be enrolled in the study once they have consented, and competed the initial assessment, and determined to meet eligibility requirements. The study team will randomize participants (N= 360) who have PTSD that is related to, has been exacerbated, or developed during the COVID-19 pandemic into CPT-Text or text-based Culturally Informed Trauma Treatment As Usual (CITT). After approximately a week of onboarding with their therapist (e.g., introduction, establishing treatment goals, etc), the active texting intervention will begin and assessments will occur at established timepoints through 24 weeks after the active intervention begins. Active interventions will occur over the course of 12 weeks. Participants will also be randomized into one of two engagement strategies: therapist reminder as usual (RAU) or RAU + incentive (RI). The study will examine an innovative incentive structure in which the study will "pay it forward" by offering free or discounted therapy to other individuals with PTSD when participants remain engaged. The study will compare the impact of an engagement strategy on treatment response and engagement, and will examine motivation as a potential mechanism. The study will also evaluate a novel Natural Language Processing (NLP) or Large-Language Model (LLM) based approach to assessing CPT-Text fidelity. This study will (1) provide critical information about how to promote sustained DMH engagement using unique incentive strategies and moderators of engagement and outcomes and (2) offer first guidance on supporting quality and fidelity of messaging-based EBTs using computational methods.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 residing in the United States
* Criterion A event measured by the Life Events Checklist for DSM-5 (LEC-5)
* Significant symptoms of PTSD as evidenced by a score of 33 or above on the PCL-5
* PTSD symptoms that began or increased during the COVID pandemic (per self-report)
* Registered/registering on Talkspace for messaging-based therapy
* Ownership of a personal device for texting
* Residence in a state with therapist capacity on the Talkspace platform

Exclusion Criteria:

* Acute risk for suicidal thoughts and/or behaviors measured by the Columbia Suicide Severity Rating Scale Lifetime-Recent Screen
* Psychosis or substance abuse that requires prioritization of treatment and/or higher level of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Baseline through 24 weeks
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that evaluates the degree to which individuals have been bothered by PTSD symptoms tied to their most currently distressing event [114] . The monthly version will be administered at baseline and the weekly version thereafter.
Engagement-Completion | 13 Weeks
  Completion of the intervention, defined as 13 weeks of CPT or CITT, or completion of all CPT modules, whichever comes first OR early completer (achievement of a PCL score below 20, which indicates good end-state functioning)

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline through 24 weeks
  The PHQ-9 [115,116] is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders that will be administered on the schedule outlined in the table. The PHQ-9 is the 9-item depression module and is a multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression.
The Brief Inventory of Psychosocial Functioning (B-IPF) | Baseline through 24 weeks
  The Brief Inventory of Psychosocial Functioning (B-IPF; [117] ) is a 7-item self-report instrument measuring respondents' level of functioning over the past 30 days in seven life domains including: romantic, family, parenting, friendship, work, education, and self-care.
The Client Satisfaction Questionnaire (CSQ) | Baseline through 24 weeks
  The Client Satisfaction Questionnaire (CSQ; [118] ) is an 8-item measure of participant satisfaction with treatment.
Working Alliance Inventory, Short Form (WAI-SF) | Week 1 through Week 12
  The Working Alliance Inventory, Short Form (WAI-SF, [125] ) is a measure to index the degree of therapeutic cohesion between the client and the therapist.
Behavioral Intention | Baseline through week 8
  Behavioral Intention (BI; which captures motivation to engage in a behavior) will be measured to examine patterns of motivation in our treatment conditions and to investigate BI as the hypothesized mechanism of change in engagement. BI measures are created based on recommendations for constructing a very brief BI measure, a frequent approach to measuring this construct, which has demonstrated reliability [119-123] . Participants will be asked, "How likely or unlikely are you to complete (baseline) or continue (mid-treatment) treatment?" on a 7-item Likert scale ranging from "Extremely Unlikely" to "Extremely Likely" at the baseline and both mid-treatment assessments.
Oppression-based traumatic stress inventory | Baseline through 24 weeks at 3 timepoints
  An assessment of trauma-related symptoms related to oppression or race/ethnicity-based trauma.
Post-traumatic Cognitions Inventory | baseline through 24 weeks, at 3 timepoints
  Assessment of common beliefs after trauma
Self-Report Altruism Scale (SRA) | Baseline
  Assessment of altruism via self-report
Cultural Humility Scale (CHS) | Week 1 through week 13, at 4 timepoints
  Assessment of important and central aspects of one's identity Assessment of customer perceptions of staff's cultural humility
Cultural Missed Opportunities (CMO) | Week 1 through week 13, at 4 timepoints
  Assessment of degree to which clients perceived that their therapist missed opportunities to discuss their cultural identity.
Engagement | 13 weeks
  THe number of days the client messaged divided by the total intervention days (days of active treatment before early response or 13 weeks, whichever comes first)
Adequate Dose of CPT | 13 weeks
  Completion of at least 8 modules of CPT-Text

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Wiltsey-Stirman, PhD, Principal Investigator — Stanford University; Katy Dondanville, PsyD, Principal Investigator — University of Texas Health Sciences Center for San Antonio
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - Talkspace LLC, New York, New York
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Investigators funded under this FOA will share those data via the National Database for Clinical Trials related to Mental Illness in a timely manner. The final quantitative dataset will be de-identified and individual records will include an NIMH Data Archive (NDA) Global Unique identifier when submitted to NDA. The research team will comply with other data submission and sharing requirements and schedule as provided in NIMH Data Archive Data Sharing Terms and Conditions (effective 7/1/15).
  Due to the sensitive nature of therapy transcripts (even when de-identified), the investigators will request explicit consent for sharing of these data but allow participants to opt out of sharing beyond the research team and institutions.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication of main outcome papers for each aim
Access Criteria: Investigators and institutions seeking data from NDA will be expected to meet data security measures, will be asked to submit a Data Use Certification co-signed by the investigator and the designated Institutional Official(s) at the NIH-recognized sponsoring institution with a current Federal Wide Assurance (FWA), and will be require to follow the procedures associated with data access described at https://ndar.nih.gov/ndarpublicweb/policies.go#sop4). Any data directly (e.g., qualitative data, outcome data) shared with other investigators would entail a data use agreement, signed by the research team and institutional authorities, and the individual(s) requesting data.

REFERENCES:
- [Background] Malgaroli M, Hull TD, Wiltsey Stirman S, Resick P. Message Delivery for the Treatment of Posttraumatic Stress Disorder: Longitudinal Observational Study of Symptom Trajectories. J Med Internet Res. 2020 Apr 29;22(4):e15587. doi: 10.2196/15587. PMID 32347814